CLINICAL TRIAL: NCT02165826
Title: A Multicenter, Randomized, Double-blind Phase 3 Study to Evaluate Tolerability and Pharmacokinetics of 500 μg Roflumilast Once Daily With an Up-titration Regimen in COPD, Including an Open-label Down-titration Period Evaluating Tolerability and Pharmacokinetics of 250 μg Roflumilast Once Daily in Subjects Not Tolerating 500 μg Roflumilast Once-daily
Brief Title: Evaluation of Tolerability and Pharmacokinetics of Roflumilast, 250μg and 500μg, as add-on to Standard COPD Treatment to Treat Severe COPD
Acronym: OPTIMIZE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RO-2455-302-RD; U1111-1150-2477 (Other: World Health Organization); 2013-001788-21 (EudraCT Number)
Record Dates: First submitted 2014-05-02; First posted 2014-06-18 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Drug therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Roflumilast 500 μg once daily (Experimental): Roflumilast 500 μg tablets, orally, once daily for 12 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive roflumilast 250 μg, tablets, orally, once daily for 8 weeks.
  Interventions: Drug: Roflumilast; Drug: Standard of Care COPD Treatment
- Roflumilast 500 μg every other day (Experimental): Roflumilast 500 μg, tablets, orally, every other day, and roflumilast placebo-matching tablets, orally, every other day on non-treatment days, for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive roflumilast 250 μg, tablets, orally, once daily for 8 weeks.
  Interventions: Drug: Roflumilast; Drug: Roflumilast Placebo; Drug: Standard of Care COPD Treatment
- Roflumilast 250 μg once daily (Experimental): Roflumilast 250 μg, tablets, orally, once daily for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive roflumilast 250 μg, tablets, orally, once daily for 8 weeks.
  Interventions: Drug: Roflumilast; Drug: Standard of Care COPD Treatment

INTERVENTIONS:
Drug: Roflumilast — Roflumilast tablets
  Other Names: Daxas, Daliresp, Libertek
Drug: Roflumilast Placebo — Roflumilast placebo-matching tablets
  Arms: Roflumilast 500 μg every other day
Drug: Standard of Care COPD Treatment — The participant is on standard of care COPD maintenance treatment including LABAs, long-acting anticholinergics, or any combination thereof taken on a constant daily dose within 12 weeks prior to Screening (Visit V0) Examples of LABA containing products are: Formoterol, Salmeterol, Indacaterol, Formoterol/Budesonide, Salmeterol/Fluticasone, Treatment including lon-acting anticholinergics: Tiotropium, Aclidinium.

SUMMARY:
The purpose of this study is to evaluate discontinuation rates of roflumilast using an up-titration regimen for the first 4 weeks of treatment compared with continuous treatment of 500 μg one daily (OD) during the entire 12-week main period, and to evaluate if participants who do not tolerate roflumilast 500 μg OD have a drug exposure with 250 μg roflumilast OD similar to that observed in other participants with the 500 μg OD dose.

DETAILED DESCRIPTION:
Roflumilast is a product which has been approved for the treatment of severe chronic obstructive lung disease (COPD) and its approved dose is 500μg once daily. This study is primarily designed to see whether alternation in this dose can improve tolerability of Roflumilast in COPD patients. Therefore one in three patients will start roflumilast therapy at a lower dose of 250μg once daily, another one in three will only take the 500μg tablet every other day (and one placebo every other day). Rest of them will start the regular dose of 500μg once daily right away and see whether starting with a lower dose of Roflumilast will lead to better tolerability. Furthermore, the study will see if patients who do not tolerate roflumilast should be given a lower dose of 250μg once daily.

Lastly, the study will investigate what the body does to roflumilast. Patients with a history of COPD for at least last 12 months and a former smoker or current smoker with history of at least 10 pack years will be invited to participate.

The main study period lasts for a maximum of 15 weeks and patients will have to visit the study site up to 6 times. If patients are not tolerating roflumilast, the investigators may switch them to the down titration period where they may be on a lower dose for rest of the study. Then patients will remain in the down titration period for additional 8 weeks and will have to visit the study site 4 times. Most of the visits will take approximately 1 to 2 hours. However, one visit in the main period and 1 or 2 visits in the down titration period will take approximately 6 to 7 hours. These visits are longer to allow time to conduct blood taking.

The Randomization visit is considered the Baseline visit and for participants that discontinue the Main Period and continue into the Down-Titration Period Day 1 of Down Titration is considered BaselineDT.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a history of chronic obstructive pulmonary disease (COPD) (according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2013) for at least 12 months prior to Screening (Visit V0) associated with chronic productive cough for 3 months in each of the 2 years prior to Screening (Visit V0, with other causes of productive cough excluded).
4. Shows a post-bronchodilator forced expiratory volume in 1 second (FEV1) of ≤50% of predicted.
5. Shows an FEV1/forced vital capacity (FVC) ratio (post-bronchodilator) <70%.
6. Has at least one documented COPD exacerbation within one year prior to Screening (Visit V0).
7. Is on standard of care COPD maintenance treatment including Long Acting β2-Agonist (LABAs), long-acting anticholinergics, or any combination thereof taken on a constant daily dose within 12 weeks prior to Screening (Visit V0).
8. Must be a former smoker (defined as smoking cessation at least one year ago) or current smoker both with a smoking history of at least 10 pack years.11
9. Is male or female and aged 40 or older.
10. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

Criteria affecting the read-out parameters of the study

1. Has a COPD exacerbation ongoing at the Screening (Visit V0), or has a COPD exacerbation between V0 and V1.
2. Has a lower respiratory tract infection not resolved 4 weeks prior to Screening (Visit V0).
3. Has a diagnosis of asthma and/or other relevant lung disease (eg, history of primary bronchiectases, cystic fibrosis, bronchiolitis, lung resection, lung cancer, interstitial lung disease [eg, fibrosis, silicosis, sarcoidosis], or active tuberculosis).
4. Has a known α1-antitrypsin deficiency.
5. Has taken roflumilast within 6 months of Screening (Visit V0).

   Criteria within ethical considerations in terms of general health
6. Has clinically relevant abnormal laboratory values suggesting an undiagnosed disease requiring further clinical evaluation (as assessed by the investigator).
7. Has a history of severe psychiatric or neurological disorders.
8. Has a history of depression associated with suicidal ideation or behavior.
9. Has congestive heart failure severity grade IV according to New York Heart Association (NYHA) Functional Classification.
10. Has hemodynamically significant cardiac arrhythmias or heart valve deformations.
11. Has computed tomography (CT) or chest x-ray findings indicating an acute pulmonary disease other than COPD (eg, tuberculosis, severe bronchiectasis, tumors).
12. Has severe immunological diseases (eg, known human immune deficiency virus (HIV) infection, multiple sclerosis, lupus erythematosus, progressive multifocal leukoencephalopathy).
13. Has liver impairment Child-Pugh B or C and/or active viral hepatitis.
14. Has severe acute infectious diseases (eg, tuberculosis, or acute hepatitis).
15. Has a history of malignant disease (except basal cell carcinoma) within 5 years before Screening (Visit V0).
16. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within one year before Screening (Visit V0).
17. Has a history of hypersensitivity or allergies to roflumilast or rescue medication or ingredients thereof, or any other contraindication for the use thereof.
18. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.
19. Intends to donate blood, organs, or bone marrow during the course of the study.
20. Has received any investigational compound within 30 days prior to Screening (Visit V0), is currently participating in another interventional clinical study, or has been previously enrolled in this study.
21. Is suspected to be unable or unwilling to comply with study procedures (eg, language problems, psychological disorders, number and timing of visits at the center).
22. Suffers from any concomitant disease that might interfere with study procedures or evaluations.
23. Is required to take excluded medications.
24. Is an immediate family member, study center employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling), or may consent under duress.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1323 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (2):
- Slovakia (2):
  - Bardejov
  - Spišská Nová Ves

REFERENCES:
- [Derived] Facius A, Marostica E, Gardiner P, Watz H, Lahu G. Pharmacokinetic and Pharmacodynamic Modelling to Characterize the Tolerability of Alternative Up-Titration Regimens of Roflumilast in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2018 Aug;57(8):1029-1038. doi: 10.1007/s40262-018-0671-4. PMID 29797235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 161 investigative sites in Bulgaria, Germany, Greece, Hungary, Korea, Philippines, Poland, Romania, Russia, Slovakia, South Africa, Spain, Thailand, Ukraine and the United Kingdom from 30 April 2014 to 21 October 2015.
Pre-assignment Details: Participants with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) were enrolled equally in 1 of 3 treatment groups in the Main Treatment Period: roflumilast 250 μg then 500 μg once daily (OD), 500 μg every other day (EOD) then 500 μg OD and 500 μg OD. Participants who discontinued received 250 μg in the Down-Titration Period.
Groups:
- Roflumilast 250 μg OD Then 500 μg OD: Roflumilast 250 μg, tablets, orally, once daily (OD) for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks in the Main Treatment Period. Any participants not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg EOD Then 500 μg OD: Roflumilast 500 μg, tablets, orally, every other day (EOD), and roflumilast placebo-matching tablets, orally, every other day on non-treatment days, for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks in the Main Treatment Period. Any participants not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg OD: Roflumilast 500 μg, tablets, orally, once daily (OD) at least 1 dose in the Main Period.
Period: Main Treatment Period
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Started | 441 | 439 | 443
Safety Analysis Set: Received Study Drug | 441 | 437 | 443
Completed | 360 | 349 | 334
Not Completed | 81 | 90 | 109
Not completed — Pre-treatment Event/Adverse Event | 44 | 57 | 68
Not completed — Major/Significant Protocol Deviation | 0 | 1 | 3
Not completed — Lost to Follow-up | 4 | 2 | 1
Not completed — Voluntary Withdrawal | 23 | 23 | 21
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Reason Not Specified | 8 | 5 | 16
Not completed — Did Not Receive Study Drug | 0 | 2 | 0
Period: Down-Titration Period
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Started | 27 | 39 | 38
Safety Analysis Set: Received Study Drug | 27 | 39 | 38
Completed | 20 | 28 | 31
Not Completed | 7 | 11 | 7
Not completed — Pre-treatment Event/Adverse Event | 4 | 10 | 3
Not completed — Voluntary Withdrawal | 2 | 1 | 2
Not completed — Reason Not Specified | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) included all randomized participants who took at least one dose of study medication. Main Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD | Total
Number analyzed (Participants) | 441 | 437 | 443 | 1321
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.81) | 65.0 (8.21) | 64.6 (8.36) | 64.6 (8.13)
Age, Customized [Number; unit: participants]
  40-64 years | 242 | 202 | 224 | 668
  65-84 years | 199 | 235 | 217 | 651
  85 years and over | 0 | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 112 | 105 | 338
  Male | 320 | 325 | 338 | 983
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 2 | 5 | 8
  Not Hispanic or Latino | 428 | 423 | 426 | 1277
  Missing | 12 | 12 | 12 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 1 | 0 | 1
  Asian | 32 | 30 | 32 | 94
  Black or African American | 3 | 3 | 3 | 9
  Native Hawaiian/Other Pacific Islander | 1 | 4 | 3 | 8
  White | 405 | 399 | 405 | 1209
Region of Enrollment [Number; unit: participants]
  Bulgaria | 36 | 18 | 30 | 84
  Germany | 12 | 24 | 16 | 52
  Greece | 8 | 6 | 6 | 20
  Hungary | 82 | 74 | 79 | 235
  Korea, Republic Of | 22 | 11 | 13 | 46
  Philippines | 7 | 13 | 10 | 30
  Poland | 60 | 68 | 71 | 199
  Romania | 54 | 46 | 44 | 144
  Russia | 37 | 48 | 55 | 140
  Slovakia | 40 | 38 | 27 | 105
  South Africa | 17 | 18 | 26 | 61
  Spain | 2 | 2 | 1 | 5
  Thailand | 2 | 6 | 9 | 17
  Ukraine | 56 | 58 | 54 | 168
  United Kingdom | 6 | 7 | 2 | 15
Height [Mean (Standard Deviation); unit: cm] | 169.1 (8.73) | 168.8 (8.66) | 169.1 (8.55) | 169.0 (8.64)
Weight [Mean (Standard Deviation); unit: kg] | 75.59 (18.627) | 74.31 (17.808) | 75.68 (16.949) | 75.20 (17.804)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.36 (5.957) | 25.98 (5.614) | 26.44 (5.888) | 26.26 (5.822)
Smoking Classification [Number; unit: participants]
  Current Smoker | 213 | 198 | 196 | 607
  Ex-smoker | 228 | 239 | 247 | 714
Number of Cigarette Pack-Years [Mean (Standard Deviation); unit: pack-years] — Number of pack-years = (number of cigarettes smoked per day/20) × number of years smoked
  pack-years | 38.1 (17.49) | 40.2 (19.22) | 37.6 (17.70) | 38.6 (18.17)
Pre-bronchodilator Forced Expiratory Volume in the First Second (FEV1) [Mean (Standard Deviation); unit: liters] | 1.022 (0.3177) | 1.028 (0.3173) | 1.018 (0.3289) | 1.023 (0.3211)
Pre-Bronchodilator Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] | 2.304 (0.7418) | 2.303 (0.7091) | 2.314 (0.6822) | 2.307 (0.7109)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Prematurely Discontinuing Study Treatment Due to Any Reason
Description: The primary endpoint is the percentage of participants prematurely discontinuing study treatment for any reason during the Main Period from Visit 1 (V1) to Last Visit (Vend). Discontinuation is defined as permanently stopping randomized treatment; participants who resume randomized treatment after an interval will not be counted as having discontinued. The analysis used discontinuations occurring during the Main Period, irrespective of whether a participant subsequently entered into the Down-Titration Period.
Time Frame: Baseline to Week 12 (Main Period)
Population: Safety Analysis Set (SAS) included all randomized participants who took at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Number analyzed (Participants) | 441 | 437 | 443
percentage of participants | 18.4 | 20.1 | 24.6
Statistical Analysis 1: Comparison: Roflumilast 250 μg OD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; p = 0.017, Regression, Logistic — Study treatment, country and baseline forced expiratory volume in the first second (FEV1) as explanatory variables; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.47 to 0.93]
Statistical Analysis 2: Comparison: Roflumilast 250 μg OD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; Cox Proportional Hazard = 0.68, 95% CI 2-sided [0.51 to 0.92] — Cox proportional hazards model with study treatment and country as class effects, and baseline FEV1 as a continuous variable
Statistical Analysis 3: Comparison: Roflumilast 500 μg EOD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; p = 0.114, Regression, Logistic — Study treatment, country and baseline forced expiratory volume in the first second (FEV1) as explanatory variables; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.55 to 1.07]
Statistical Analysis 4: Comparison: Roflumilast 500 μg EOD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; Cox Proportional Hazard = 0.77, 95% CI 2-sided [0.58 to 1.02] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With Adverse Events of Interest
Description: Adverse events of interest to evaluate tolerability are defined as diarrhea, nausea, headache, decreased appetite, insomnia and abdominal pain.
Time Frame: Baseline to Week 12 (Main Period)
Population: SAS included all randomized participants who took at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Number analyzed (Participants) | 441 | 437 | 443
percentage of participants | 45.4 | 48.3 | 54.2
Statistical Analysis 1: Comparison: Roflumilast 250 μg OD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; p = 0.001, Regression, Logistic — Study treatment, country and baseline forced expiratory volume in the first second (FEV1) as explanatory variables; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.47 to 0.83]
Statistical Analysis 2: Comparison: Roflumilast 500 μg EOD Then 500 μg OD vs Roflumilast 500 μg OD; Analyses were performed using a hierarchical testing procedure; Test type: Superiority or Other; p = 0.091, Regression, Logistic — Study treatment, country and baseline forced expiratory volume in the first second (FEV1) as explanatory variables; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.59 to 1.04]

3. Secondary Outcome: Change From Baseline (V0DT) in Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1) to Final Visit of the Down-Titration Period
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using spirometry prior to taking study medication A positive change from Baseline indicates improvement.
Time Frame: Baseline (V0DT) [assessment at end of main period] and Final Visit of Down-Titration Period (Up to Day 56)
Population: Participants from the Down-Titration Period Full Analysis Set (FAS), all randomized participants who entered this period, regardless of whether they took study medication, with data available for analysis.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period: Participants in the roflumilast 250 μg once daily (OD) then 500 μg OD who were not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg EOD_Down-Titration Period: Participants in the roflumilast 500 μg, every other day (EOD) treatment arm who were not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg OD_Down Titration Period: Participants in the roflumilast 500 μg once daily (OD) treatment arm who were not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Number analyzed (Participants) | 26 | 39 | 38
Liters | 0.030 (0.2294) | 0.055 (0.4170) | 0.007 (0.3555)

4. Secondary Outcome: Percentage of Participants Prematurely Discontinuing Study Treatment Due to Any Reason During Down-Titration Period
Time Frame: Baseline DT (Day 1 of Down-Titration Period) to Week 8 (Down-Titration Period)
Population: Down-Titration Period Full Analysis Set (FAS) included all randomized participants who entered this period, regardless of whether they took study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Number analyzed (Participants) | 27 | 39 | 38
percentage of participants | 25.9 | 28.2 | 18.4

5. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1) During the Down-Titration Period
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using spirometry prior to taking study medication. A positive change from Baseline indicates improvement.
Time Frame: Baseline DT (Day 1 of Down-Titration Period) to Days 14, 28 and 56 (Down-Titration Period)
Population: Down-Titration Period Full Analysis Set (FAS) included all randomized participants who entered this period, regardless of whether they took study medication. "n" in each category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Number analyzed (Participants) | 27 | 39 | 38
Liters
  Day 14 (n=20, 32, 34) | 0.128 (0.3708) | 0.223 (0.4101) | 0.097 (0.2532)
  Day 28 (n=20, 29, 31) | 0.162 (0.4274) | 0.218 (0.4443) | 0.070 (0.2067)
  Day 56 (n=26, 39, 38) | 0.162 (0.3311) | 0.261 (0.4616) | 0.127 (0.3334)

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1) During the Main Period
Description: as for outcome 5
Time Frame: Baseline (Day 1 of Main Period) to Days 15, 29, 57 and 84 (Main Period)
Population: Main Period FAS included all randomized participants, regardless of whether they took study medication. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Number analyzed (Participants) | 441 | 439 | 443
Liters
  Day 15 (n=409, 406, 386) | 0.067 (0.2299) | 0.094 (0.2573) | 0.094 (0.2566)
  Day 29 (n=402, 389, 365) | 0.099 (0.2605) | 0.115 (0.2629) | 0.116 (0.2440)
  Day 57 (n=376, 367, 352) | 0.104 (0.2659) | 0.161 (0.2765) | 0.133 (0.2705)
  Day 84 (n=402, 411, 409) | 0.117 (0.2690) | 0.141 (0.2882) | 0.122 (0.2705)

7. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Vital Capacity (FVC) During the Main Period
Description: Forced vital capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Pulmonary function testing was performed using spirometry prior to taking study medication. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1 of Main Period) to Days 15, 29, 57 and 84 (Main Period)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Number analyzed (Participants) | 441 | 439 | 443
Liters
  Day 15 (n=409, 406, 386) | 0.096 (0.4053) | 0.112 (0.4168) | 0.104 (0.4166)
  Day 29 (n=402, 389, 365) | 0.139 (0.3826) | 0.143 (0.4172) | 0.149 (0.4173)
  Day 57 (n=376, 367, 352) | 0.156 (0.4346) | 0.194 (0.4974) | 0.162 (0.4341)
  Day 84 (n=402, 411, 409) | 0.157 (0.4746) | 0.207 (0.4925) | 0.147 (0.4555)

8. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Vital Capacity (FVC) During the Down-Titration Period
Description: as for outcome 7
Time Frame: Baseline DT (Day 1 of Down-Titration Period) to Days 14, 28 and 56 (Down-Titration Period)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Number analyzed (Participants) | 27 | 39 | 38
Liters
  Day 14 (n=20, 32, 34) | 0.087 (0.5392) | 0.303 (0.5103) | 0.104 (0.4568)
  Day 28 (n=20, 29, 31) | 0.125 (0.6151) | 0.191 (0.4780) | 0.067 (0.3522)
  Day 56 (n=26, 39, 38) | 0.167 (0.5492) | 0.113 (0.5100) | 0.029 (0.4628)

9. Secondary Outcome: Change From Baseline in Treatment Satisfaction Scores During the Main Period
Description: Participants will be asked to assess their satisfaction with their COPD therapy at each visit. The participants will rate their treatment satisfaction on a 7-point scale where 0=very satisfied, 1=satisfied, 2=somewhat satisfied, 3=neither satisfied nor dissatisfied, 4=somewhat dissatisfied, 5=dissatisfied and 6=very dissatisfied. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1 of Main Period) to Days 15, 29, 57 and 84 (Main Period)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD | Roflumilast 500 μg EOD Then 500 μg OD | Roflumilast 500 μg OD
Number analyzed (Participants) | 441 | 439 | 443
score on a scale
  Day 15 (n=410, 408, 386) | -0.4 (1.12) | -0.3 (1.15) | -0.3 (1.07)
  Day 29 (n=403, 390, 366) | -0.5 (1.23) | -0.5 (1.16) | -0.5 (1.22)
  Day 57 (n=375, 369, 351) | -0.6 (1.24) | -0.6 (1.26) | -0.5 (1.29)
  Day 84 (n=407, 416, 412) | -0.5 (1.43) | -0.5 (1.51) | -0.3 (1.52)

10. Secondary Outcome: Change From Baseline in Treatment Satisfaction Scores During the Down-Titration Period
Description: as for outcome 9
Time Frame: Baseline DT (Day 1 of Down-Titration Period) to Days 14, 28 and 56 (Down-Titration Period)
Population: Down-Titration Period Full Analysis Set (FAS) included all randomized participants who entered this period, regardless of whether they took study medication. "n" in each of the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Number analyzed (Participants) | 27 | 39 | 38
score on a scale
  Day 14 (n=20, 32, 34) | -1.1 (1.85) | -0.8 (1.57) | -0.8 (1.84)
  Day 28 (n=20, 29, 31) | -1.2 (2.01) | -0.8 (1.75) | -0.9 (1.81)
  Day 56 (n=26, 39, 38) | -0.8 (2.23) | -0.3 (2.15) | -0.4 (2.26)

11. Secondary Outcome: Population PK Model Point Estimate for Absorption Rate Constant (Ka) of Roflumilast and Roflumilast N-oxide
Description: PK model point estimates for Ka are calculated using all available PK data for all doses of roflumilast combined and are presented for roflumilast and metabolite roflumilast N-oxide. Results are reported for the subgroups defined according to the covariates (weight, age, smoking status and sex) included in the final model.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours at weeks 2 or 8
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration.
Measure: Number; unit: units per hour (1/h)
Groups:
- All PK Participants_Roflumilast: All PK participants who received any dose of roflumilast. Results for roflumilast.
- All PK Participants_Roflumilast N-oxide: All PK participants who received any dose of rofumilast. Results for roflumilast N-oxide.
Arm/Group | All PK Participants_Roflumilast | All PK Participants_Roflumilast N-oxide
Number analyzed (Participants) | 1238 | 1238
units per hour (1/h)
  Weight=33.5 kg | 0.90 | 0.57
  Weight=70 kg | 0.90 | 0.57
  Weight=160 kg | 0.90 | 0.57
  Age=40 | 0.90 | 0.57
  Age=60 | 0.90 | 0.57
  Age=92 | 0.90 | 0.57
  Smoking=former | 0.90 | 0.57
  Smoking=current | 0.90 | 0.57
  Sex=female | 0.90 | 0.57
  Sex=male | 0.90 | 0.57

12. Secondary Outcome: Population PK Model Point Estimate for Apparent Oral Clearance (CL/F) of Roflumilast and Roflumilast N-oxide
Description: PK model point estimates for CL/F are calculated using all available PK data for all doses of roflumilast combined and are presented for roflumilast and metabolite roflumilast N-oxide. Results are reported for the subgroups defined according to the covariates (weight, age, smoking status and sex) included in the final model.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours at weeks 2 or 8
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration.
Measure: Number; unit: liters per hour (L/h)
Arm/Group | All PK Participants_Roflumilast | All PK Participants_Roflumilast N-oxide
Number analyzed (Participants) | 1238 | 1238
liters per hour (L/h)
  Weight=33.5 kg | 5.64 | 0.73
  Weight=70 kg | 5.64 | 0.89
  Weight=160 kg | 5.64 | 1.12
  Age=40 | 7.23 | 1.11
  Age=60 | 5.64 | 0.89
  Age=92 | 4.35 | 0.71
  Smoking=former | 5.64 | 0.89
  Smoking=current | 6.50 | 1.03
  Sex=female | 5.64 | 0.89
  Sex=male | 5.64 | 0.79

13. Secondary Outcome: Population PK Model Point Estimate for Apparent Central Volume (Vc/F) of Roflumilast and Roflumilast N-oxide
Description: PK model point estimates for Vc/F are calculated using all available PK data for all doses of roflumilast combined and are presented for roflumilast and metabolite roflumilast N-oxide. Results are reported for the subgroups defined according to the covariates (weight, age, smoking status and sex) included in the final model.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours at weeks 2 or 8
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration.
Measure: Number; unit: liters (L)
Arm/Group | All PK Participants_Roflumilast | All PK Participants_Roflumilast N-oxide
Number analyzed (Participants) | 1238 | 1238
liters (L)
  Weight=33.5 kg | 26.0 | 4.5
  Weight=70 kg | 63.9 | 11.0
  Weight=160 kg | 175.2 | 30.2
  Age=40 | 63.9 | 11.0
  Age=60 | 63.9 | 11.0
  Age=92 | 63.9 | 11.0
  Smoking=former | 63.9 | 11.0
  Smoking=current | 63.9 | 11.0
  Sex=female | 63.9 | 11.0
  Sex=male | 63.9 | 11.0

14. Secondary Outcome: Population PK Model Point Estimate for Apparent Peripheral Volume (Vp/F) of Roflumilast and Roflumilast N-oxide
Description: PK model point estimates for Vp/F are calculated using all available PK data for all doses of roflumilast combined and are presented for roflumilast and metabolite roflumilast N-oxide. Results are reported for the subgroups defined according to the covariates (weight, age, smoking status and sex) included in the final model.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours at weeks 2 or 8
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration.
Measure: Number; unit: L
Arm/Group | All PK Participants_Roflumilast | All PK Participants_Roflumilast N-oxide
Number analyzed (Participants) | 1238 | 1238
L
  Weight=33.5 kg | 69.6 | 5.0
  Weight=70 kg | 171.0 | 12.4
  Weight=160 kg | 468.8 | 34.0
  Age=40 | 171.0 | 12.4
  Age=60 | 171.0 | 12.4
  Age=92 | 171.0 | 12.4
  Smoking=former | 171.0 | 12.4
  Smoking=current | 171.0 | 12.4
  Sex=female | 171.0 | 12.4
  Sex=male | 171.0 | 12.4

15. Secondary Outcome: Total PDE4 Inhibitory Activity (tPDE4i)
Description: tPDE4i was derived using in-vitro constants for protein binding and biochemical activity (IC50). tPDE4i is reported for a set of reference participants defined according to the covariates included in the final model.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours post-dose at Days 15 and 57. Down-titration: Pre-dose and 1,2,3,4,6 hours post-dose at Days 1 and 14 and pre-dose at Days 28 and 56.
Population: Participants from the PK Set, all participants who had at least 1 quantifiable PK concentration, with data available. Study design only includes the 250 µg arm for analyses of this outcome measure in the Down-Titration period. Measured values are predicted values reported as median and 90% prediction interval.
Measure: Median (90% Confidence Interval); unit: unitless
Groups:
- Roflumilast 500 μg EOD: Roflumilast 500 μg, tablets, orally, every other day (EOD) in the Main Period.
- Roflumilast 250 μg OD: Roflumilast 250 μg tablets, orally, once daily in the Main Period.
- Roflumilast 250 µg Down-Titration: 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
Arm/Group | Roflumilast 500 μg OD | Roflumilast 500 μg EOD | Roflumilast 250 μg OD | Roflumilast 250 µg Down-Titration
Number analyzed (Participants) | 392 | 399 | 404 | 101
unitless
  Overall | 1.17 [0.366 to 2.05] | 0.608 [0.227 to 1.03] | 0.563 [0.157 to 1.01] | 0.583 [0.210 to 1.24]
  Age < 65 (n=198,187,229,45) | 1.06 [0.323 to 1.85] | 0.559 [0.237 to 0.998] | 0.518 [0.160 to 0.958] | 0.511 [0.205 to 0.984]
  Age ≥ 65 to < 75 (n=146,159,136,39) | 1.24 [0.550 to 2.08] | 0.660 [0.177 to 1.04] | 0.614 [0.138 to 1.10] | 0.683 [0.207 to 1.23]
  Age ≥ 75 (n=48,53,39,17) | 1.24 [0.318 to 2.31] | 0.676 [0.188 to 1.12] | 0.616 [0.195 to 1.01] | 0.712 [0.300 to 1.32]
  Weight < 60 kg (n=56,78,73,17) | 1.34 [0.591 to 2.64] | 0.755 [0.258 to 1.22] | 0.653 [0.156 to 1.12] | 0.934 [0.325 to 1.39]
  Weight ≥ 60 kg (n=336,321,331,84) | 1.12 [0.339 to 1.99] | 0.592 [0.223 to 1.01] | 0.552 [0.158 to 0.971] | 0.538 [0.202 to 1.02]
  Males (n=300,297,290,66) | 1.12 [0.363 to 1.96] | 0.585 [0.226 to 0.994] | 0.558 [0.145 to 0.998] | 0.575 [0.213 to 1.14]
  Females (n=92,102,114,35) | 1.29 [0.468 to 2.38] | 0.696 [0.260 to 1.15] | 0.618 [0.189 to 1.01] | 0.626 [0.217 to 1.25]
  Current Smoker (n=179,183,200,45) | 1.04 [0.327 to 1.88] | 0.568 [0.247 to 0.976] | 0.514 [0.101 to 0.949] | 0.554 [0.228 to 1.21]
  Former Smoker (n=213,216,204,56) | 1.25 [0.416 to 2.15] | 0.632 [0.186 to 1.09] | 0.626 [0.196 to 1.10] | 0.624 [0.207 to 1.30]

16. Secondary Outcome: Summary Statistics of Predicted Total PDE4 Inhibitory Activity (tPDE4i)
Description: tPDE4i was derived using in-vitro constants for protein binding and biochemical activity (IC50). An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. Adverse Events of Interest (AEI) for PK analyses included: headache, diarrhea, nausea, vomiting, abdominal pain, appetite disorders, sleep disorders, angioedema, psychiatric disorders (anxiety, nervousness), psychiatric disorders (depression,suicidal ideation,behaviour) and weight loss.
Time Frame: as for outcome 15
Population: PK Set included all participants who had at least 1 quantifiable PK concentration. "n" in the category is the number of participants with available data. Study design only includes the 250 µg OD and 500 µg OD arms for analyses of this outcome measure. Measured values are predicted values reported as median and 90% prediction interval.
Measure: Median (90% Confidence Interval); unit: unitless
Groups:
- Roflumilast 250 μg OD: Roflumilast 500 μg at least one dose in the Main Period followed by Roflumilast 250 μg tablets, orally, once daily in the Down -Titration Period.
Arm/Group | Roflumilast 500 μg OD | Roflumilast 250 μg OD
Number analyzed (Participants) | 1114 | 76
unitless
  All Participants (n=1114,76) | 1.17 [0.352 to 2.03] | 0.611 [0.197 to 1.243]
  Discontinuation due to Any AEI=Yes (n=67,62) | 1.28 [0.427 to 2.22] | 0.647 [0.201 to 1.239]
  Discontinuation due to Any AEI=No (n=1047,14) | 1.16 [0.339 to 2.02] | 0.436 [0.212 to 1.069]
  Discontinuation due to Any AE=Yes (n=77,64) | 1.29 [0.464 to 2.10] | 0.647 [0.204 to 1.237]
  Discontinuation due to Any AE=No (n=1037,12) | 1.16 [0.337 to 2.02] | 0.408 [0.209 to 1.006]
  Discontinuation Due to Any Reason=Yes (n=106,75) | 1.23 [0.416 to 2.06] | 0.600 [0.197 to 1.243]
  Discontinuation Due to Any Reason=No (n=1008,1) | 1.16 [0.332 to 2.02] | 0.626 [0.626 to 0.626]
  At Least 1 AEI=Yes (n=536,75) | 1.23 [0.453 to 2.09] | 0.600 [0.197 to 1.243]
  At Least 1 AEI=No (578,1) | 1.12 [0.297 to 1.98] | 0.929 [0.929 to 0.929]
  At Least 1 AE=Yes (n=693,76) | 1.22 [0.416 to 2.07] | 0.611 [0.197 to 1.243]
  At Least 1 AE=No (n=421,0) | 1.08 [0.294 to 1.97] | NA [NA to NA] — No participants in this category for this arm.

17. Secondary Outcome: Median Simulated Percentage of Participants With Adverse Events of Interest
Description: The PK model predicted the total PDE4 inhibitory activity and the median simulated percentage of participants with Adverse Events of Interest during 12 weeks of treatment based on 1000 participants simulated. Results are reported for the set of reference participants defined according to the covariates [weight, smoking status, sex, age and long acting muscarinic antagonist (LAMA)] included in the final model and tPDE4i. Adverse Events of Interest (AEI) for PK analyses included: headache, diarrhea, nausea, vomiting, abdominal pain, appetite disorders, sleep disorders, angioedema, psychiatric disorders (anxiety, nervousness), psychiatric disorders (depression, suicidal ideation, behaviour) and weight loss.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours post-dose at Days 15 and 57. AEIs: 12 Weeks
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration. Number of participants analyzed is the number of participants simulated. Measured values are predicted values.
Measure: Number; unit: percentage of participants
Groups:
- Roflumilast 250 μg OD: Roflumilast 250 μg, tablets, orally, once daily (OD) at least 1 dose in the Main Period.
- Roflumilast 500 μg EOD: Roflumilast 500 μg, orally, every other day (EOD) at least 1 dose in the Main Period
Arm/Group | Roflumilast 250 μg OD | Roflumilast 500 μg EOD | Roflumilast 500 μg OD
Number analyzed (Participants) | 1000 | 1000 | 1000
percentage of participants
  Weight=48 kg (tPDE4i=0.72,0.72,1.45) | 53.2 [0.352 to 2.03] | 53.2 [0.197 to 1.243] | 61.8
  Weight=74 kg (tPDE4i=0.65,0.65,1.30) | 52.3 [0.427 to 2.22] | 52.3 [0.201 to 1.239] | 60.1
  Weight=105 kg (tPDE4i=0.60.0.60,1.19) | 51.7 [0.339 to 2.02] | 51.7 [0.212 to 1.069] | 58.8
  Former Smoker (tPDE4i=0.65,0.65,1.30) | 52.3 [0.464 to 2.10] | 52.3 [0.204 to 1.237] | 60.1
  Current Smoker (tPDE4i=0.56,0.56,1.13) | 42.5 [0.337 to 2.02] | 42.5 [0.209 to 1.006] | 49.2
  Male (tPDE4i=0.65,0.65,1.30) | 52.3 [0.416 to 2.06] | 52.3 [0.197 to 1.243] | 60.1
  Female (tPDE4i=0.72,0.72,1.45) | 53.2 [0.332 to 2.02] | 53.2 [0.626 to 0.626] | 61.8
  Age=51 (tPDE4i=0.58,0.58,1.15) | 51.4 [0.453 to 2.09] | 51.4 [0.197 to 1.243] | 58.4
  Age=64 (tPDE4i=0.65,0.65,1.30) | 52.3 [0.297 to 1.98] | 52.3 [0.929 to 0.929] | 60.1
  Age=77 (tPDE4i=0.72,0.72,1.44) | 53.2 [0.416 to 2.07] | 53.2 [0.197 to 1.243] | 61.7
  With LAMA (tPDE4i=0.65,0.65,1.30) | 52.3 [0.294 to 1.97] | 52.3 [NA to NA] | 60.1
  Without LAMA (tPDE4i=0.65,0.65,1.30) | 43.5 | 43.5 | 51.4

18. Secondary Outcome: Median Simulated Absolute Change From Baseline in FEV1 at Weeks 4 and 12
Description: The PK model predicted the total PDE4 inhibitory activity and the median simulated Change from Baseline (CFB) in FEV1 at Week 4 and the Change from Baseline in FEV1 at Week 12 during 12 weeks of treatment with roflumilast 500 μg OD based on 1000 participants simulated. Results are reported for the set of reference participants defined according to the covariates [weight, smoking status, sex, age, race, COPD severity, concomitant long acting muscarinic antagonist (LAMA) and Percent FEV1 reversibility] included in the final model and tPDE4i. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing was performed using spirometry prior to taking study medication. A positive change from Baseline indicates improvement.
Time Frame: Main period: Pre-dose and 1,2,3,4,6 hours post-dose or pre-dose and 2 hours post-dose at Days 15 and 57. FEV-1: Pre-dose and Weeks 4 and 12
Population: Pharmacokinetic (PK) Set included all participants who had at least 1 quantifiable PK concentration. The number of participants analyzed is the number of participants simulated. Measured values are predicted values.
Measure: Number; unit: milliliters (mL)
Groups:
- Roflumilast 500 μg OD_CFB in FEV1 @ Week 4: Roflumilast 500 μg, tablets, orally, once daily (OD) for 12 weeks. Results for Change from Baseline in FEV1 at Week 4.
- Roflumilast 500 μg OD_CFB in FEV1 @ Week 12: Roflumilast 500 μg, tablets, orally, once daily (OD) for 12 weeks. Results for Change from Baseline in FEV1 at Week 12.
Arm/Group | Roflumilast 500 μg OD_CFB in FEV1 @ Week 4 | Roflumilast 500 μg OD_CFB in FEV1 @ Week 12
Number analyzed (Participants) | 1000 | 1000
milliliters (mL)
  Weight=33.5 kg (tPDE4i=1.012,1.012) | 50 [0.197 to 1.243] | 32
  Weight=70 kg (tPDE4i=0.839,0.839) | 60.5 [0.201 to 1.239] | 56
  Weight=160 kg (tPDE4i=0.681,0.681) | 108 [0.212 to 1.069] | 157
  Current Smoker (tPDE4i=0.729,0.729) | 99.5 [0.204 to 1.237] | 96.5
  Former/Never Smoker (tPDE4i=0.839,0.839) | 60.5 [0.209 to 1.006] | 56
  Male (tPDE4i=0.839,0.839) | 60.5 [0.197 to 1.243] | 56
  Female (tPDE4i=0.937,0.937) | 53.2 [0.626 to 0.626] | 49.8
  Age=40 years (tPDE4i=0.675,0.675) | 57.6 [0.197 to 1.243] | 52.2
  Age=60 years (tPDE4i=0.839,0.839) | 60.5 [0.929 to 0.929] | 56
  Age=92 years (tPDE4i=1.06,1.06) | 56.4 [0.197 to 1.243] | 53.3
  Asian (tPDE4i=0.839,0.839) | 56.1 [NA to NA] | 52
  non-Asian (tPDE4i=0.839,0.839) | 60.5 | 56
  COPD_Not Very Severe (tPDE4i=0.839,0.839) | 60.5 | 56
  COPD_Very Severe (tPDE4i=0.839,0.839) | 42.2 | 39.1
  LAMA=Yes (tPDE4i=0.839,0.839) | 60.5 | 56
  LAMA=No (tPDE4i=0.839,0.839) | 63.5 | 58.8
  %FEV1 Reversibility=-28% (tPDE4i=0.839,0.839) | 68.1 | 63.1
  %FEV1 Reversibility=10% (tPDE4i=0.839,0.839) | 60.5 | 56
  %FEV1 Reversibility=147% (tPDE4i=0.839,0.839) | 32.9 | 30.5

ADVERSE EVENTS:
Time Frame: Main Treatment Period: First dose of study drug to 30 days past last dose or first dose in the Down-Titration Period (Up to 114 Days). Down-Titration Period: First dose of study drug to 30 days past the last dose of study drug (Up to 86 Days).
Description: Due to the design of the study, the most common (≥ 2%) non-serious adverse events were determined separately for each period, the blinded Main Treatment Period and the open-label Down-Titration Period. A result of 0 means that the event did not meet the ≥ 2% threshold for that study period but did meet the threshold for the other study period.
Groups:
- Roflumilast 250 μg OD Then 500 μg OD_Main Treatment Period: Roflumilast 250 μg, tablets, orally, once daily (OD) for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks in the Main Treatment Period. Any participants not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg EOD Then 500 μg OD_Main Treatment Period: Roflumilast 500 μg, tablets, orally, every other day (EOD), and roflumilast placebo-matching tablets, orally, every other day on non-treatment days, for 4 weeks, followed by roflumilast 500 μg, tablets, orally, once daily, for 8 weeks in the Main Treatment Period. Any participants not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
- Roflumilast 500 μg OD_Main Treatment Period: Roflumilast 500 μg tablets, orally, once daily for 12 weeks in the Main Treatment Period. Any participants not tolerating study treatment were prematurely discontinued and received roflumilast 250 μg, tablets, orally, once daily for 8 weeks in the open-label Down-Titration Period.
Arm/Group | Roflumilast 250 μg OD Then 500 μg OD_Main Treatment Period | Roflumilast 500 μg EOD Then 500 μg OD_Main Treatment Period | Roflumilast 500 μg OD_Main Treatment Period | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period | Roflumilast 500 μg EOD_Down-Titration Period | Roflumilast 500 μg OD_Down Titration Period
Serious Adverse Events (participants affected / at risk) | 19/441 | 22/437 | 20/443 | 1/27 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 239/441 | 248/437 | 272/443 | 13/27 | 21/39 | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 250 μg OD Then 500 μg OD_Main Treatment Period (N=441) | Roflumilast 500 μg EOD Then 500 μg OD_Main Treatment Period (N=437) | Roflumilast 500 μg OD_Main Treatment Period (N=443) | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period (N=27) | Roflumilast 500 μg EOD_Down-Titration Period (N=39) | Roflumilast 500 μg OD_Down Titration Period (N=38)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 500 μg OD and is not related (previous AE included severe syncope).
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 250 μg OD then 500 μg OD and is not related (previous AE included moderate COPD).
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 250 μg OD then 500 μg OD and is not related (previous AE included moderate COPD).
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 500 μg OD and is not related (previous AE included concurrent moderate haemoptysis).
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 13 | 7 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 250 μg OD then 500 μg OD and is not related (previous AE included concurrent moderate pneumonia).
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with roflumilast 500 µg EOD then 500 µg OD and is not related.
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast 250 μg OD Then 500 μg OD_Main Treatment Period (N=441) | Roflumilast 500 μg EOD Then 500 μg OD_Main Treatment Period (N=437) | Roflumilast 500 μg OD_Main Treatment Period (N=443) | Roflumilast 250 μg OD Then 500 μg OD_Down Titration Period (N=27) | Roflumilast 500 μg EOD_Down-Titration Period (N=39) | Roflumilast 500 μg OD_Down Titration Period (N=38)
Diarrhoea (Gastrointestinal disorders) | 107 | 113 | 134 | 3 | 6 | 11
Nausea (Gastrointestinal disorders) | 87 | 92 | 110 | 1 | 5 | 8
Abdominal pain (Gastrointestinal disorders) | 69 | 58 | 64 | 0 | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 19 | 15 | 27 | 0 | 3 | 3
Fatigue (General disorders) | 4 | 10 | 5 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 11 | 12 | 0 | 0 | 3
Weight decreased (Investigations) | 10 | 9 | 17 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 100 | 105 | 129 | 3 | 8 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 21 | 20 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7 | 9 | 0 | 0 | 0
Headache (Nervous system disorders) | 107 | 115 | 115 | 2 | 7 | 10
Dizziness (Nervous system disorders) | 16 | 20 | 14 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 97 | 100 | 106 | 2 | 10 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 34 | 39 | 38 | 3 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 13 | 11 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 6 | 4 | 9 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.